CLINICAL TRIAL: NCT04111055
Title: Feasibility of Computer-assisted Vasopressor Infusion Using Continuous Noninvasive Blood Pressure Monitoring in High-risk Patients Undergoing Renal Transplant Surgery
Brief Title: Closed-loop Vasopressor Infusion Using Continuous Noninvasive Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018-276
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Hemodynamic (MAP) Stability

STUDY DESIGN:
Intervention Model Description: Single prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop group (Experimental): The MAP of the patient will be managed by the CLV system to avoid hypotension. The MAP target selected in the closed-loop system will be the patient's MAP target ( same target as patient's MAP value preoperatively). Then the closed-loop system will have to adjust norepinephrine infusion rate to keep that MAP value within 10% of patient's target.
  Interventions: Device: Closed-loop system

INTERVENTIONS:
Device: Closed-loop system — the CLV system will correct hypotension by automated adjustment of norepinephrine.

SUMMARY:
Intraoperative hypotension and blood pressure variability are associated with postoperative complications in surgical patients.

The investigators have developed a closed-loop vasopressor (CLV) controller that titrates norepinephrine to correct hypotension.

After having tested the system in a small cohort series of patients undergoing major surgeries, the investigators aimed to test the feasibility of the CLV controller guided noninvasively and continuously with the ClearSight system (Edwards Lifesciences, USA) in three high risk patients undergoing renal transplant surgery

DETAILED DESCRIPTION:
Intraoperative hypotension is frequent in patients undergoing surgery and can negatively impact organ perfusion.

The investigators have developed a closed-loop vasopressor (CLV) controller to more efficiently correct hypotension.

The investigators tested it extensively in preclinical studies and recently demonstrated its feasibility and excellent performance metrics in a short series of high-risk patients undergoing major surgical procedures.

In these studies, the controller was linked to a minimally-invasive advanced hemodynamic monitoring device utilizing an arterial line which then controlled a vasopressor infusion. However, the vast majority of patients who undergo surgery do not require an arterial line but should still benefit from rapid corrections of hypotensive episodes that are less rapidly detected via an intermittent non-invasive blood pressure cuff. Fortunately, completely noninvasive technology now allows us to continuously monitor blood pressure and therefore extend the use of our closed-loop vasopressor system to patients in whom an arterial catheter would not typically be placed. Patients undergoing renal transplant surgeries are the ideal patient population.

The investigators aimed to test the feasibility of guiding our CLV controller with a continuous noninvasive blood pressure monitoring device (ClearSight system, Edwards Lifesciences, Irvine, CA, USA) in three patients (case series)

ELIGIBILITY:
Inclusion Criteria:

1. Adult high risk patients undergoing renal transplant surgery
2. Patients equipped with a clearsight advanced hemodynamic monitoring system

Exclusion Criteria:

1. Atrial fibrillation
2. No consent obtained from the patient.
3. Ejection fraction < 30%

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Percentage of case time in hypotension | during surgery
  % of case time without hypotension. MAP of at least 5mmHg below the chosen CLV target

SECONDARY OUTCOMES:
Percentage of active treatment time spent in a hypertensive state | during surgery
  Percentage of active treatment time spent in a hypertensive state, defined as a MAP >5mmHg above the chosen target MAP with an active norepinephrine infusion
Amount of vasopressor used | during surgery
  Amount of vasopressor administered to the patient
Incidence of acute kidney injury | 30 days postsurgery
  Incidence of acute kidney injury defined with the KDIGO classification

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre J Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No